CLINICAL TRIAL: NCT04500366
Title: GERAS Frailty Rehabilitation at Home: Virtual Bundled Care for Seniors Who Are Frail to Build Strength and Resilience During COVID-19
Brief Title: GERAS Frailty Rehabilitation at Home During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Director, GERAS Centre for Aging Research, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11408
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Frailty
Keywords: Rehabilitation; Frailty; COVID-19; Exercise; Protein; Medication
MeSH Terms: conditions — Frailty; COVID-19; Motor Activity | interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two arms (35/arm based on sample size calculation) for 12-weeks of socialization only or multi-modal frailty rehabilitation. The socialization only arm will receive 1x/week phone calls from medical student volunteers. Multi-modal frailty rehabilitation will involve virtual care including 1x/week socialization, 2x/week exercise (small group physiotherapy live-streamed sessions), nutrition (virtual consult), and medication support (virtual pharmacist consult) all via a videoconferencing service.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors, the study biostatistician, the investigative team, and the steering committee will be blinded to intervention assignments. Research assistants, study intervention personnel (pharmacist, instructors) and participants will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socialization (Active Comparator): Participants randomized to the socialization arm will receive once-weekly phone calls from medical student volunteers for a total of 12-weeks (n=35). This program pairs health professional student volunteers with older adults in the community to provide social comfort while heightened physical distancing measures are in place during the current COVID-19 pandemic. Attendance and duration of the phone calls will be logged.
  Interventions: Behavioral: Socialization
- Multi-Modal Frailty Rehabilitation (Experimental): Multi-modal frailty rehabilitation will involve virtual care including 1x/week socialization, 2x/week exercise (small group physiotherapy live-streamed sessions), nutrition (virtual consult), and medication support (virtual pharmacist consult) all through a videoconferencing system.
  Interventions: Behavioral: Socialization; Behavioral: Virtual Group Exercise; Combination Product: Nutrition Consult and Protein Supplementation; Behavioral: Medication Review

INTERVENTIONS:
Behavioral: Socialization — Social interaction is associated with better mental and physical health, and evidence suggests that group versus individual engagement may offer unique cognitive benefits for older adults as well as peer reinforcement and encouragement.
Behavioral: Virtual Group Exercise — Participants will receive twice-weekly (one hour per class) virtual exercise via small-group physiotherapy sessions for a total of 12 weeks. All exercise sessions will occur virtually via a videoconferencing system. The classes will focus on functional movements specifically designed for seniors with frailty and mobility challenges, and will include modifications for gait aids such as canes or walkers. Class sizes will be small to allow for tailoring of exercises based on challenging, safe, progressive, evidence-based exercises. In accordance with recent guidelines to achieve 3 hours/week for fall prevention practice in older adults, participants will also be provided with tailored supplemental home exercises developed by the study physiotherapist to gain an additional 1 hour of physical activity.
  Arms: Multi-Modal Frailty Rehabilitation
Combination Product: Nutrition Consult and Protein Supplementation — Nutrition Consult: Participants will be scheduled for a one-on-one virtual nutrition consult. During the consultation, study staff will assess the nutritional status of the participant and will provide them with counselling and coaching to improve their nutrition.
  Protein Supplementation: Oral nutrition supplements commercially available from Nestle will be provided unless contraindicated. The oral nutrition supplement contains 360 calories and 14 grams of protein per serving. Participants are advised to take this with a meal or within 3 hours of exercise on activity days.
  Arms: Multi-Modal Frailty Rehabilitation
Behavioral: Medication Review — A study pharmacist will review the participant's medication list and will utilize Beers and/or START/STOPP criteria to provide recommendations to optimize/update their medications to the participant's healthcare provider. Study geriatricians will be listed as contacts on the primary care provider recommendations and available for consultation.
  Arms: Multi-Modal Frailty Rehabilitation

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic is keeping people apart, which can take a toll on physical and mental health. Many healthcare professionals are concerned vulnerable seniors may become deconditioned, which substantially increases risk of health complications and need for hospitalization. To address the immediate impact of COVID-19 policies (i.e., physical distancing, reduced access to care), the GERAS Frailty Rehabilitation model will be adapted to be delivered remotely in the homes of vulnerable seniors. The investigators' aim is to understand how to best build resilience among vulnerable seniors in the community through at-home rehabilitation services (socialization, exercise, nutrition, and medication support).

DETAILED DESCRIPTION:
During this unprecedented time of COVID-19, many healthcare professionals are concerned that vulnerable seniors who are housebound and isolated will become deconditioned resulting in functional losses in mental status, continence and ability to complete activities of daily living. Total inactivity in seniors can result in a 10-20% decrease in muscle strength per week (1 -3% per day). Loss of muscle strength may quickly convert a vulnerable older adult who was ambulatory into a bedridden state. This will affect the health of seniors and increase demand on healthcare systems. An innovative model to deliver frailty rehabilitation services remotely is urgently needed to: 1) increase access to specialized services 2) provide added supports for seniors discharged from the hospital who are in need of rehabilitation and 3) build resilience in seniors to prevent re-hospitalization or institutionalization. Therefore, to address the immediate impact of COVID-19 policies (i.e., physical distancing and reduced access to care), the GERAS Frailty Rehabilitation model will be adapted to be delivered remotely in the homes of vulnerable seniors. This proof-of-concept, randomized control trial aims to understand how to best build resilience among vulnerable seniors through at-home rehabilitation services using socialization, exercise, nutrition, and medication support.

The short-term immediate goals for this RCT are to help vulnerable seniors who are isolated because of physical distancing measures to build strength and resilience throughout the COVID-19 pandemic. The major deliverables are 1) the adaptation of an in-person program to virtual delivery 2) the piloting of a care pathway with inter-disciplinary professionals that can be expanded to reach a larger number of individuals.

The long-term goal of the study is the seamless implementation of a new model for multimodal Frailty Rehabilitation that closes the care gap in rehabilitation for frail seniors in the immediate and foreseeable future.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged ≥ 65 years of age;
* Score between 4-6 (inclusive) on the clinical frailty scale;
* Able to ambulate independently with or without a walking aid; OR with caregiver supervision at home;
* Obtain clearance for exercise: For hospital referrals - average resting heart rate between 50-100 bpm and average blood pressure less than or equal to 160/90mmHg (as per Canadian Society for Exercise Physiology guidelines for exercise clearance); OR Self- referrals: Obtain exercise clearance from their family physician prior to the first intervention session.

Exclusion Criteria:

* Unable to speak or understand English and has no caregiver for translation;
* Significant cognitive impairment where they may have difficulty following two-step commands;
* Receiving palliative/end of life care;
* Unstable angina or unstable heart failure;
* Travel plans that would result in missing greater than 20% of the trial's 12-week duration;
* Currently attending a group exercise program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Physical Function | Baseline and 12 Weeks Post-Intervention
  Assessed by the 5x Sit-to-Stand (time to complete). Faster times to complete indicate better performance.
Change in Mental Health | Baseline and 12 Weeks Post-Intervention
  Assessed by the Depression Anxiety Stress Scale (DASS-21). Higher scores indicate greater risk of depression, anxiety and stress [depression, anxiety, stress subscores range 0-21].

SECONDARY OUTCOMES:
Change in Sarcopenia | Baseline and 12 Weeks Post-Intervention
  Assessed by the SARC-F - Self-reported strength, assistance with walking, rising from a chair, climbing stairs and falls. Higher scores indicate greater level of sarcopenia [range 0-10].
Change in Frailty | Baseline and 12 Weeks Post-Intervention
  Assessed by the Fit-Frailty Index. Higher scores indicate greater degree of frailty [range 0-1].
Change in Self-Efficacy | Baseline and 12 Weeks Post-Intervention
  Balance confidence will be assessed using the Activities-specific Balance Confidence Scale (ABCs). Higher scores indicate greater balance confidence [range 0-100].
Self-Reported Change in Function, Health and Well-Being | Baseline and 12 Weeks Post-Intervention
  Assessed by the interRAI Community Rehab Assessment - Self-Report
Clinician-Reported Change in Function, Health and Well-Being | Baseline and 12 Weeks Post-Intervention
  Assessed by the interRAI Community Rehab Assessment - Clinician-Completed
Change in Fitness | Weekly up to 12 weeks
  Assessed by the Borg Rate of Perceived Exertion after exercise. Higher scores indicate greater level of exertion [range 6-20]. Also assessed using accelerometers (heart rate, sedentary time, physical activity time, energy expenditure).
Program Satisfaction | 12 Weeks Post-Intervention
  Assessed using a program questionnaire in accordance with the Kirkpatrick 5-Level Evaluation Model. Scores will be on a 5-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree".
Change in Health-Related Quality of Life | Baseline and 12 Weeks Post-Intervention
  Assessed by the EQ-5D-5L scale. Lower scores indicate better self-reported quality of life [range 0-100].
Change in Nutrition | Baseline and 12 Weeks Post-Intervention
  Assessed by the Subjective Global Assessment. Grades range from A-C where 'A' represents normal nutrition and 'C' represents severe malnourishment.
Change in Emergency Room Visits | Baseline and 12 Weeks Post-Intervention
  Number of emergency room visits will be recorded. Higher number of emergency room visits indicates higher healthcare utilization.
Change in Hospitalizations | Baseline and 12 Weeks Post-Intervention
  Number of hospitalizations will be recorded. Higher number of hospitalizations indicates higher healthcare utilization.
Change in Number of Calls to 911 | Baseline and 12 Weeks Post-Intervention
  Number of calls to 911 will be recorded. Higher number of calls indicates higher healthcare utilization.

OTHER OUTCOMES:
Feasibility Outcome #1 - Reach of intervention | 12 Weeks Post-Intervention
  Assessed by the number of individuals who participated. Target reach is 70 participants.
Feasibility Outcome #2 - Adoption of the Intervention | 12 Weeks Post-Intervention
  Assessed by number of referral sites. Target is 5 referral sites.
Feasibility Outcome #3 - Implementation of the Intervention | 12 Weeks Post-Intervention
  Assessed by the number of individuals who completed the intervention. Higher number of individuals completing the study indicates greater success in implementation.
Feasibility Outcome #4 - Maintenance of the Intervention | 12 Weeks Post-Intervention
  Assessed by the number of referral sites continuing with a second cohort. Greater number of referral sites continuing with a second cohort indicates greater maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, Principal Investigator — Scientific Director, GERAS Centre for Aging Research
Locations (1):
- McMaster University - Hamilton Health Sciences (St. Peter's Site), Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Okpara C, Ioannidis G, Thabane L, Adachi JD, Rabinovich A, Hewston P, Lee J, McArthur C, Kennedy C, Woo T, Boulos P, Bobba R, Wang M, Thrall S, Mangin D, Marr S, Armstrong D, Patterson C, Bray S, de Wit K, Maharaj S, Misiaszek B, Sookhoo JB, Thompson K, Papaioannou A. The Geras virtual frailty rehabilitation program to build resilience in older adults with frailty during COVID-19: a randomized feasibility trial. Pilot Feasibility Stud. 2023 Jul 17;9(1):124. doi: 10.1186/s40814-023-01346-7. PMID 37461117